CLINICAL TRIAL: NCT01045720
Title: The Treatment Effect of 2 Traditional Chinese Medicines[Suo Quan Wan]and [Wu Lin San] in Clozapine-induced Hypersalivation in Schizophrenia Patient.
Brief Title: The Treatment of 2 Chinese Medicines in Clozapine-induced Hypersalivation in Schizophrenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: IRB TCVGH, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C08200
Record Dates: First submitted 2010-01-05; First posted 2010-01-11 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Schizophrenia; Clozapine; Hypersalivation; Traditional Chinese Medicine
Keywords: Schizophrenia; clozapine; hypersalivation; Suo Quan Wan; Wu Lin San
MeSH Terms: conditions — Schizophrenia; Sialorrhea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Placebo
- ChinesMed (Experimental)
  Interventions: Drug: Suo Quan Wan, Wu Lin San

INTERVENTIONS:
Drug: Suo Quan Wan, Wu Lin San — Suo Quan Wan Wu Lin San Placebo 2/daily
  Arms: ChinesMed
Drug: Placebo — Placebo (starch)
  Arms: Placebo Comparator

SUMMARY:
The goal of this research is hoping to combine traditional Chinese medicine medication and find out how to solve clozapine-induced hypersalivation, also reduce side-effect, medication compliance, improving life quality, improving social-function and reducing neopathy.

DETAILED DESCRIPTION:
Clozapine, an antipsychotic drug, is an important clinical medicine which is used for schizophrenia and preventing for its relapse; clozapine is better than some other atypical antipsychotics. However, in clinical uses, clozapine often could induce hypersalivation, it is not only influencing patient's appearance, also deteriorating sleeping quality which could deter patient discontinuing to take medicine.

In previous researches, Suo Quan Wan and Wu Lin San had been proven effective for hypersalivation and no significant side-effects, nevertheless, it still lack of systematical scientific trial reports. The ingredients of Suo Quan Wan are Wu Yao, San Yao and Yi Zhi Ren; the ingredients of Wu Lin San are Gui Zhi, Fu Ling, Zhu Ling, Ze Xie and Bai Ju, both have bi-directional regulatory functions for body fluid and saliva.

The goal of this research is hoping to combine traditional Chinese medicine medication and find out how to solve clozapine-induced hypersalivation, also reduce side-effect, medication compliance, improving life quality, improving social-function and reducing neopathy.

ELIGIBILITY:
Inclusion Criteria:

1.20 year and older. All genders. 2.Psychiatry doctor diagnosed schizophrenia or schizoaffective disorder will be recruited for participation in this study.

3.Using clozapine as an antipsychotic drug and has a side-effect of hypersalivation.

4.Testee agree and sign informed consent forms to do this experiment.

Exclusion Criteria:

1. Use clozapine as an antipsychotic drug not over 8 weeks.
2. Testee have other diseases could influence saliva secretion, such as Parkinson's disease.
3. Pregnant, prepare to pregnant within half a year or in the lactation period.
4. Add or alter following medicines within 2 weeks:

   4.1 Central acting 2-adrenergic receptor agonist 4.2 anticholinergic/antimuscarinic drugs 4.3 b-adrenoreceptor blockers, diphenhydramine, botulinum toxin injection
5. Testee's lever function test (AST/ALT) is higher than 3 (4 weeks medication).
6. Testee's kidney function test (Cr) is higher than 2.5mg/dl (4 weeks medication).
7. Testee have participate other medicine trial within one month.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tsuo-Hung Lan, MD., PhD., Study Director — Taichung Veterans General Hospital; Tsuo-Hung Lan, MD.,PhD, Study Director — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan, Taiwan

REFERENCES:
- [Derived] Hung CC, Fu PK, Wang HY, Chan CH, Lan TH. Treatment effects of traditional Chinese medicines Suoquan Pill and Wuling Powder on clozapine-induced hypersalivation in patients with schizophrenia: study protocol of a randomized, placebo-controlled trial. Zhong Xi Yi Jie He Xue Bao. 2011 May;9(5):495-502. PMID 21565135